CLINICAL TRIAL: NCT06915337
Title: GI Windows Flexagon Self Forming Magnet Anastomosis Plus OTOLoc for Creating Gastric-Jejunal Anastomoses in Patients Undergoing Surgical Procedures
Brief Title: Magnet Anastomosis in Patients Undergoing Gastric Surgery
Acronym: MAPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIW 25-002
Record Dates: First submitted 2025-04-02; First posted 2025-04-08 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Gastric Anastomosis (Site)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Study Group: Prospective Evaluation of Flexagon SFM Device with OTOLoc (Experimental): This is a multicenter, single-arm study in which clinical outcomes are prospectively evaluated for subjects undergoing gastric-jejunal anastomosis using the Flexagon SFM Device with OTOLoc.
  Interventions: Device: Gastric-Jejunal Anastomosis with Flexagon SFM Device with OTOLoc

INTERVENTIONS:
Device: Gastric-Jejunal Anastomosis with Flexagon SFM Device with OTOLoc — This study will investigate one type of intervention: gastric-jejunal anastomosis creation in subjects undergoing surgical procedures. Flexagon SFMs and OTOLoc devices will be delivered laparoscopically and/or endoscopically into portions of the stomach and the jejunum that are intended to be anastomosed. An OTOLoc device will be deployed into the gastric wall of the stomach to provide access for the deployment of a Flexagon SFM into the stomach. The process is repeated at an intended section of jejunum. Once deployed, the Flexagon SFMs are approximated and positioned, after which the SFMs are couple together to form the anastomosis, with the OTOLoc devices allowing fluidic communication between the two lumens until the anastomosis is fully formed.

SUMMARY:
The primary objective of this trial is to investigate the safety and effectiveness of the Flexagon SFM system plus OTOLoc when used to create a gastro-jejunal anastomosis in participants undergoing gastric surgery.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm clinical study to evaluate the GI Windows Flexagon Self Forming Magnet Anastomosis plus OTOLoc for creating gastric-jejunal anastomoses in patients undergoing gastric surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 22 years or older at screening
2. Candidate for gastric surgery requiring gastro-jejunal or gastro-ileal anastomosis with cardiac/medical clearance for surgery
3. Able to understand and sign informed consent document
4. American Society of Anesthesiologists (ASA) score < IV at time of procedure
5. Lives, and intends to remain, within a 300 kilometers radius of study center for the duration of the study
6. Able to refrain from smoking during study follow-up period

Exclusion Criteria:

1. Known or suspected allergy to silicone, nickel, titanium or Nitinol
2. BMI > 55 kg/m2
3. Uncontrolled diabetes (defined as HbA1c >10%)
4. Congenital or acquired anomalies of the GI tract, including atresia or malrotation that would inhibit passing of SFM magnet
5. Diagnosed with obstructed or perforated colon cancer
6. Any documented conditions for which endoscopy and/or laparoscopy would be contraindicated or history of previous technically difficult or failed endoscopy
7. Any previous major surgery on the stomach, duodenum, hepatobiliary tree (excluding laparoscopically removed gallbladder or prior sleeve gastrectomy), pancreas or right colon
8. Coagulation deficiency not normalized by medical treatment or platelet count <50,000/µL
9. Known moderate to severe renal disease (eGFR < 44 milliliters per minute per 1.73m2) or ongoing dialysis
10. Hyperkalemia / hypercoagulability or prior Venus Thromboembolism / Pulmonary Embolism
11. Immunocompromised (e.g., active treatment for malignancies, hematologic malignancy, on immunosuppressive therapy, moderate or severe primary immunodeficiency, advanced or untreated HIV, active treatment with high-dose corticosteroids (i.e., 20 or more mg of prednisone or equivalent per day when administered for 2 or more weeks prior to surgery) or other immunosuppressive or immunomodulatory agents
12. Active H. pylori infection Participants with active H. pylori may continue with the screening process if they are treated via medication
13. Active or suspected infection at the surgical site or a CDC Class 3/contaminated or Class 4/dirty-infected surgical wound.
14. Obstructive Sleep Apnea on CPAP unless assessed and cleared by independent physician
15. Contraindication to general anesthesia
16. Breast-feeding, pregnant, or planning on becoming pregnant during the follow-up period
17. Currently participating or has participated in another clinical trial within the past 30 days and is receiving/has received an investigational drug, device, or biologic agent
18. Participant is not appropriate for inclusion in the clinical trial, per the medical opinion of the Principal Investigator

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Successful Anastomosis Creation without the Need for Reoperation | 30 Days
  The study's primary endpoint (patient success) is defined as successful anastomosis created with the Flexagon SFM without placement procedure, device or target anastomosis-related reoperation through 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD, Principal Investigator — Bhandari Hospital & Research Centre; Pablo Marin, MD, Principal Investigator — Clinica Colonial Hospital
Locations (2):
- Clinica Colonial Hospital, Santiago, Huechuraba, Región Metropolitana, Chile
- Mohak Hitech Specialty Hospital, Indore, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.